CLINICAL TRIAL: NCT05521555
Title: Return to Work After Total Knee Arthroplasty in Patients Under 55, a Retrospective Study in an University Hospital
Brief Title: Return to Work After Total Knee Arthroplasty in Young Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Didier MAINARD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2022-A00947-36
Record Dates: First submitted 2022-08-23; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Knee Arthritis
Keywords: total knee arthroplasty; return to work; arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- total knee arthroplasty under 55: Patient who had total knee arthroplasty before 55 between January 2010 and December 2019
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — First intention total knee arthroplasty

SUMMARY:
This study takes its base in the augmenting number of primary total knee arthroplasty in the world whom quality and survey had permit to widen their indications to younger patients who are in the age of professional activity.

This work will focus on young patients under 55 who had had primary total knee arthroplasty, retrospectively, over the past 10 years, to determine the factors influencing early or late return to work, depending of socio economics factors.

This will optimize the information for the patient, and prepare him if necessary for a long work stop, and possibly obtain a better satisfaction for him.

DETAILED DESCRIPTION:
The primary aim of this study is to determine the rate of young patients returning to work after a primary total knee arthroplasty and the mean delay, and to compare it to other studies.

The mean delay of return to work in the literature is between 8 to 12 weeks, with up to 98% of patients returning to work.

The investigators will next determine which category of patients could have a late return to work superior to 6 months, and also if the surgery could give back a professional activity to patients who were in a long work stoppage.

ELIGIBILITY:
Inclusion Criteria:

* first intention total knee arthroplasty
* Age at the time of surgery under 55

Exclusion Criteria:

* Not in capacity of completing a questionnaire
* revision of total knee arthroplasty

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who underwent a total knee arthroplasty, under 55 at the time of surgery, with or without professional activity at the time of surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Return to work in weeks | 2 years
  Duration between surgery and return to work

CONTACTS AND LOCATIONS:
Overall Officials: Didier MAINARD, PHD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Hopital central, Nancy, Meurthe Et Moselle, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: return to work after total knee or hip arthroplasty — https://pubmed.ncbi.nlm.nih.gov/34863957/